CLINICAL TRIAL: NCT01213277
Title: Differences in Hemoglobin Glycation Rate in Diabete Mellitus Patients
Brief Title: A1c Discordance in Diabetes Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: a pilot study of 7 patients did not reveal a temperature dependent difference in glycation rates
Sponsor: Endocrine Research Society (Other)
Responsible Party: Dr. Hugh Tildesley, Providence Health Care
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: A1c Discordance
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; HbA1c; Glycation Rate; Fructosamine
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast Glycator (Active Comparator): The subjects enrolled in this study will have a fructosamine test and blood drawn to see whether they are fast glycators
  Interventions: Other: Fast Glycator
- Control (Active Comparator): These patients will have their blood drawn to know what the normal glycation rate is in diabetic patients
  Interventions: Other: Control

INTERVENTIONS:
Other: Fast Glycator — The subjects enrolled in this study will have a fructosamine test and blood drawn to see whether they are fast glycators
  Arms: Fast Glycator
Other: Control — These patients will have their blood drawn to know what the normal glycation rate is in diabetic patients
  Arms: Control

SUMMARY:
HbA1c is used as a gold standard to see whether patients have optimal glycemic control. Today, many physicians rely solely on HbA1c to change medication. However, there is a select group of patients that have low average glucose levels but high HbA1c levels. The investigators believe that these patients are fast glycators meaning that they incorporate sugar into their hemoglobin faster than normal. The investigators want to determine whether these patients are fast glycators.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diabetes
* Patients who test their sugar levels at least 3 times daily
* Recorded diary of sugar levels for the past month
* Willingness to have blood drawn
* Willingness to allow their blood sugar diary to be photocopied
* Estimated average glucose as derived from A1c is ≥ 4 mmol from measured glucose from self-monitoring blood glucose testing

Exclusion Criteria:

* Patient with medical conditions that may affect their study participation or results will be excluded.
* Patients who are anemic
* Renal insufficient with a serum creatinine level > 200 μmol/L

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-05

PRIMARY OUTCOMES:
Primary endpoint is to see whether they are fast glycators | One Week

SECONDARY OUTCOMES:
A secondary endpoint includes adverse events such as unplanned hospitalizations for any cause that last more than 24 hours | One Week

REFERENCES:
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Cohen RM, Holmes YR, Chenier TC, Joiner CH. Discordance between HbA1c and fructosamine: evidence for a glycosylation gap and its relation to diabetic nephropathy. Diabetes Care. 2003 Jan;26(1):163-7. doi: 10.2337/diacare.26.1.163. PMID 12502674
- [Background] Hempe JM, Gomez R, McCarter RJ Jr, Chalew SA. High and low hemoglobin glycation phenotypes in type 1 diabetes: a challenge for interpretation of glycemic control. J Diabetes Complications. 2002 Sep-Oct;16(5):313-20. doi: 10.1016/s1056-8727(01)00227-6. PMID 12200073
- [Background] McCarter RJ, Hempe JM, Gomez R, Chalew SA. Biological variation in HbA1c predicts risk of retinopathy and nephropathy in type 1 diabetes. Diabetes Care. 2004 Jun;27(6):1259-64. doi: 10.2337/diacare.27.6.1259. PMID 15161772
- [Background] Gould BJ, Davie SJ, Yudkin JS. Investigation of the mechanism underlying the variability of glycated haemoglobin in non-diabetic subjects not related to glycaemia. Clin Chim Acta. 1997 Apr 4;260(1):49-64. doi: 10.1016/s0009-8981(96)06508-4. PMID 9101100